CLINICAL TRIAL: NCT06690385
Title: Registry of Patients Included in the DEPRECAP (Lung Cancer Screening Porgramme by Low-dose Computed Tomography for Patients With Chronic Obstructive Pulmonary Disease (COPD) or Emphysema.
Brief Title: DEPRECAP: Lung Cancer Screening Programme by LDCT for Patients With COPD or Emphysema.
Acronym: DEPRECAP
Status: Recruiting | Type: Observational
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Principal Investigator, Carolina Maria Gotera Rivera, Pneumologist, Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Other Study IDs: ER2_EO180-19_FJD-HGV
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer; COPD; Emphysema
Keywords: Lung cancer screening; Low-dose computed CT; COPD; Emphysema
MeSH Terms: conditions — Lung Neoplasms; Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 40 Years
Biospecimen Retention: Samples Without DNA — Biological samples: serum, plasma and whole blood obtained at inclusion and during follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD or Emphysema: COPD according to GOLD guidelines determined by spirometry or pulmonary emphysema on previous chest CT or by CO diffusion test values less than 80%.

SUMMARY:
The DEPRECAP (Early detection of lung cancer) study is an ongoing, prospective, longitudinal, multicenter lung cancer screening program that recruited individuals with COPD or emphysema from the pulmonary clinics of Fundación Jiménez Díaz University Hospital and Villalba General Hospital, in Madrid, Spain.

The aim of this observational study is to determine the scientific evidence needed to study the benefit and potential effects of lung cancer screening in this group of patients and to determine the long-term effects of the intervention in reducing the high mortality rates associated with late-stage lung cancer diagnosis in a very high-risk population, to address under-diagnosis of COPD and to promote smoking cessation. This leads to the creation of a registry with clinical, radiological, functional data and biological samples for future studies in this cohort of patients to provide the scientific evidence needed to study the benefit and potential effects of screening for lung cancer and other tobacco-related pathologies diagnosed by Low-dose CT (LDCT)

DETAILED DESCRIPTION:
Participants who met the inclusion/exclusion criteria detailed below and agreed to participate, underwent annual LDCT and pulmonary function tests until age 75 or 15 years of smoking abstinence, whichever came first. The study protocol was approved by the Ethics Committee of the Fundación Jiménez Díaz (ER2_EO180-19_FJD-HGV) and all participants signed their informed consent.

Inclusion criteria were males or females, 55-75 years of age, current or former smokers (Less than 15 years of abstinence) with a cumulative smoking exposure of greather than 30 pack-years and a diagnosis of COPD according to the GOLD guidelines and/or emphysema identified by LDCT. Individuals with a recent history of cancer (except non-melanoma skin cancer or carcinoma in situ) as well as those with other medical conditions that posed a significant risk of death were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Current or former smokers (>15 years of abstinence) with a cumulative smoking exposure of > 30 pack-years
* Diagnosis of COPD according to the GOLD guidelines and/or emphysema identified by LDCT and/or a carbon monoxide diffusing capacity (DLCO) lower than 80% of predicted (as per the Global Lung Function Initiative (GLI) equations)

Exclusion Criteria:

* Individuals with a recent history of cancer (except non-melanoma skin cancer or carcinoma in situ) as well as those with other medical conditions that posed a significant risk of death were excluded from the study.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All those patients who agree to be part of the DEPRECAP programme registry corresponding to the reference population of the Fundación Jiménez Díaz and General de Villalba hospitals in the Community of Madrid (Spain).
Sampling Method: Non-Probability Sample
Enrollment: 1998 (Estimated)
Dates: Start 2014-01-14 (Actual); Primary Completion 2024-11-13 (Estimated); Study Completion 2024-11-13 (Estimated)

PRIMARY OUTCOMES:
Lung cancer screening | 15 years
  Creation of a multi-centre pilot lung cancer screening programme targeting high-risk subjects.
  with COPD and emphysema.

SECONDARY OUTCOMES:
Lung cancer screening | 15 years
  To create a multicenter registry of clinical data, radiological images and blood samples to provide scientific evidence to study the benefit of lung cancer screening in patients with COPD or emphysema.
Lung cancer screening: smoking cessation | 15 years
  To determine the effect of primary and secondary prevention on smoking cessation as a key element in the follow-up of the patients included.

OTHER OUTCOMES:
Lung cancer screening: comorbidities associated | 15 years
  Use follow-up in the screening programme to diagnose high-impact comorbidities associated with smoking such as COPD, pulmonary emphysema, bronchiectasis, incipient interstitial lung disease (ILA) or established interstitial lung disease and coronary heart disease.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Gotera, MD, Principal Investigator — Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Locations (2):
- Spain (2):
  - Fundación Jimenez Díaz Universitary Hospital, Madrid
  - Pneumology department. Fundación Jimenez Díaz University Hospital, Madrid

IPD SHARING:
Plan to Share IPD: No
I haven't decided at the moment.